CLINICAL TRIAL: NCT05007054
Title: Long-Term Outcomes of Different Treatment Strategies in Patients With Three-Vessel Coronary Disease
Brief Title: Long-Term Outcomes in Patients With Three-Vessel Disease
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: YJ-KY-FB-2021-10
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Three Vessel Coronary Disease
Keywords: three-vessel coronary disease; percutaneous coronary intervention; coronary artery bypass grafting; medical therapy; clincial outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Percutaneous coronary intervention: The PCI performed following current standard guidelines. All patients were pre-treated with aspirin and clopidogrel before catheterization. Thereafter, heparin (70-100 IU/kg) was administered before PCI, however, the use of glycoprotein IIb/IIIa inhibitors was at the physician's discretion. Dual-antiplatelet medication was administered to the patients after PCI for at least 12 months.
  Interventions: Procedure: PCI or CABG
- Coronary artery bypass grafting: The left internal mammary artery was routinely used to graft to the left anterior descending artery and completed by venous grafts to other coronary branches with standard bypass techniques. Te procedure was performed by surgeons experienced in onpump or of-pump surgery at the operator's discretion.
  Interventions: Procedure: PCI or CABG
- Medical therapy: Patients with neither PCI nor CABG treatment were allocated to the MT alone group. For medical therapy, antiplatelet medication, statins, renin-angiotensin system blockade, β-blockers, and nitrate were used.

INTERVENTIONS:
Procedure: PCI or CABG — The PCI performed following current standard guidelines. All patients were pre-treated with aspirin and clopidogrel before catheterization. Thereafter, heparin (70-100 IU/kg) was administered before PCI, however, the use of glycoprotein IIb/IIIa inhibitors was at the physician's discretion. Dual-antiplatelet medication was administered to the patients after PCI for at least 12 months. For CABG, the left internal mammary artery was routinely used to graft to the left anterior descending artery and completed by venous grafts to other coronary branches with standard bypass techniques. The procedure was performed by surgeons experienced in on-pump or of-pump surgery at the operator's discretion.
  Groups: Coronary artery bypass grafting; Percutaneous coronary intervention

SUMMARY:
The long-term outcome of coronary artery bypass grafting (CABG), percutaneous coronary intervention (PCI), and medical therapy (MT) alone for triple-vessel disease (TVD) patients is controversial. The aim of this study is to evaluate the long-term outcome of TVD patients among these three treatment strategies, to find out the most appropriate treatment methods for these patients.

DETAILED DESCRIPTION:
The present study was a retrospective observational study. Patients who underwent diagnostic coronary angiography from January 2013 to December 2018 were eligible for this study if they had three-vessel disease, which was defined as more than 50% stenosis in three major epicardial coronary arteries, left anterior descending, left circumﬂex, and right coronary artery. There were no pre-specified exclusion criteria. The choice of PCI, CABG, or MT was mainly followed the guidelines and based on clinical and angiographic features, physical condition (comorbidities, malignant tumor, frailty, etc.), complexity, and was discussed by physicians and surgeons, combined with the choice of patients. The PCI strategy and stent type were left to the physician's discretion.

The primary endpoint were major adverse cardiac and cerebrovascular events (MACCE), which were a composite of all-cause death, myocardial infarction (MI), repeat revascularization, or stroke. Clinical information of in-hospital outcome was obtained by reviewing medical records. Follow-up was completed by survey via telephone, letter, or hospital visit. All patients had at least one follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed as having three-vessel disease (defined as angiographic stenosis of ≥ 50% in all three main epicardial coronary arteries, with or without left main artery involvement) and age >18 years.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with three-vessel coronary disease.
Sampling Method: Probability Sample
Enrollment: 4300 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | The median follow-up time was 2.4 years.
  MACCEs were a composite of all-cause death, myocardial infarction (MI), repeat revascularization, or stroke.

SECONDARY OUTCOMES:
Cardiac death, MI, repeat revascularization, stroke, or hospitalization for angina pectoris or heart failure | The median follow-up time was 2.4 years.
  Cardiac death was considered to be of cardiac origin cause could be established. MI was defined as recurrent symptoms with new electrocardiographic changes compatible with MI or cardiac markers at least twice the upper limit of normal. Repeat revascularization was defined as either PCI or CABG in the vessel for any reasons. Stroke was defined as ischemic or hemorrhagic stroke either occurring during hospitalization or requiring hospitalization for symptoms. Hospitalization for angina pectoris or heart failure heart failure was defined as hospitalization because of worsening angina pectoris or heart failure requiring intravenous drug therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Guo, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

REFERENCES:
- [Result] Escaned J, Collet C, Ryan N, De Maria GL, Walsh S, Sabate M, Davies J, Lesiak M, Moreno R, Cruz-Gonzalez I, Hoole SP, Ej West N, Piek JJ, Zaman A, Fath-Ordoubadi F, Stables RH, Appleby C, van Mieghem N, van Geuns RJ, Uren N, Zueco J, Buszman P, Iniguez A, Goicolea J, Hildick-Smith D, Ochala A, Dudek D, Hanratty C, Cavalcante R, Kappetein AP, Taggart DP, van Es GA, Morel MA, de Vries T, Onuma Y, Farooq V, Serruys PW, Banning AP. Clinical outcomes of state-of-the-art percutaneous coronary revascularization in patients with de novo three vessel disease: 1-year results of the SYNTAX II study. Eur Heart J. 2017 Nov 7;38(42):3124-3134. doi: 10.1093/eurheartj/ehx512. PMID 29020367
- [Result] Mohr FW, Morice MC, Kappetein AP, Feldman TE, Stahle E, Colombo A, Mack MJ, Holmes DR Jr, Morel MA, Van Dyck N, Houle VM, Dawkins KD, Serruys PW. Coronary artery bypass graft surgery versus percutaneous coronary intervention in patients with three-vessel disease and left main coronary disease: 5-year follow-up of the randomised, clinical SYNTAX trial. Lancet. 2013 Feb 23;381(9867):629-38. doi: 10.1016/S0140-6736(13)60141-5. PMID 23439102
- [Result] Head SJ, Davierwala PM, Serruys PW, Redwood SR, Colombo A, Mack MJ, Morice MC, Holmes DR Jr, Feldman TE, Stahle E, Underwood P, Dawkins KD, Kappetein AP, Mohr FW. Coronary artery bypass grafting vs. percutaneous coronary intervention for patients with three-vessel disease: final five-year follow-up of the SYNTAX trial. Eur Heart J. 2014 Oct 21;35(40):2821-30. doi: 10.1093/eurheartj/ehu213. Epub 2014 May 21. PMID 24849105
- [Result] Shiomi H, Morimoto T, Furukawa Y, Nakagawa Y, Tazaki J, Sakata R, Okabayashi H, Hanyu M, Shimamoto M, Nishiwaki N, Komiya T, Kimura T; CREDO-Kyoto PCI/CABG Registry Cohort-2 Investigators. Comparison of Five-Year Outcome of Percutaneous Coronary Intervention With Coronary Artery Bypass Grafting in Triple-Vessel Coronary Artery Disease (from the Coronary Revascularization Demonstrating Outcome Study in Kyoto PCI/CABG Registry Cohort-2). Am J Cardiol. 2015 Jul 1;116(1):59-65. doi: 10.1016/j.amjcard.2015.03.040. Epub 2015 Apr 7. PMID 25956622
- [Result] Xu JJ, Zhang Y, Jiang L, Tian J, Song L, Gao Z, Feng XX, Zhao XY, Zhao YY, Wang D, Sun K, Xu LJ, Liu R, Gao RL, Xu B, Song L, Yuan JQ. Comparison of Long-term Outcomes in Patients with Premature Triple-vessel Coronary Disease Undergoing Three Different Treatment Strategies: A Prospective Cohort Study. Chin Med J (Engl). 2018 Jan 5;131(1):1-9. doi: 10.4103/0366-6999.221273. PMID 29271373
- [Result] Zhao X, Xu L, Jiang L, Tian J, Zhang Y, Wang D, Sun K, Xu B, Zhao W, Hui R, Gao R, Song L, Yuan J. Real-world outcomes of different treatment strategies in patients with diabetes and three-vessel coronary disease: a mean follow-up 6.3 years study from China. Cardiovasc Diabetol. 2021 Jan 11;20(1):16. doi: 10.1186/s12933-020-01193-3. PMID 33430864
- [Result] Tsuneyoshi H, Komiya T, Kadota K, Shimamoto T, Sakai J, Hiraoka T, Wada K, Kaneko H, Fujimoto Y, Furuichi Y, Hata R, Jinno T, Tominaga O. Coronary artery bypass surgery is superior to second generation drug-eluting stents in three-vessel coronary artery disease: a propensity score matched analysis. Eur J Cardiothorac Surg. 2017 Sep 1;52(3):462-468. doi: 10.1093/ejcts/ezx031. PMID 28874027